CLINICAL TRIAL: NCT04967196
Title: Phase 1 Study of the Administration of Ipilimumab Intra-Lymphatically Using the Sofusa® DoseConnect™ DEVICE With Nivolumab Administered IV in Patients With Metastatic Melanoma
Brief Title: Ipilimumab and Nivolumab for the Treatment of Stage III-IV Unresectable Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC200711; NCI-2021-06866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-013238 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (ipilimumab DC and IV, nivolumab) CLOSED (Experimental): Patients receive ipilimumab intra-lymphatically via DoseConnect™ on day 1 of cycle 1 and IV over 30 minutes on day 1 of cycles 2-4. Patients also receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo lymphatic imaging with ICG prior to treatment start and blood sample collection throughout the study. (CLOSED TO ENROLLMENT)
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Procedure: Lymph Node Assessment; Procedure: Biospecimen Collection
- Cohort B (Ipilimumab DC and nivolumab IV) (Experimental): Patients receive ipilimumab intra-lymphatically via DoseConnect™ and nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study and may optionally undergo lymphatic imaging with ICG prior to treatment start.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Procedure: Lymph Node Assessment; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Ipilimumab — Given via DoseConnect device or IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Procedure: Lymph Node Assessment — Undergo lymphatic imaging with ICG
  Other Names: Lymph Node Examination
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I trial identifies the best dose of ipilimumab that can be administered through the DoseConnect™ device followed by nivolumab in treating patients with stage III melanoma that cannot be removed by surgery (unresectable) or stage IV melanoma that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of ipilimumab that can be administered through the DoseConnect™ device followed 30 minutes later by nivolumab intravenously (IV) on day 1 of a 21-day cycle in patients with metastatic melanoma. (Cohort A) II. To determine the maximum tolerated dose (MTD) of ipilimumab that can be administered through up to four (4) DoseConnect™ devices, followed by nivolumab IV on Day 1 of four 21-day cycle in patients with metastatic melanoma. (Cohort B)

SECONDARY OBJECTIVE:

I. To assess the pharmacokinetics of ipilimumab administered using the DoseConnect™ followed by nivolumab IV in patients with metastatic melanoma. (Cohort A) II. To assess the rate of Grade 3 and 4 adverse events, as well as the rate of drug discontinuation for adverse events and objective response rate (ORR) for patients who receive ipilimumab via the DoseConnect™ device for four cycles in combination with nivolumab administered as an IV infusion, without any IV administration of ipilimumab. (Cohort B)

CORRELATIVE OBJECTIVE:

I. To assess the changes in immunologic profile after one cycle of ipilimumab administered using the DoseConnect™ followed by nivolumab IV.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive ipilimumab intra-lymphatically via DoseConnect™ on day 1 of cycle 1 and IV over 30 minutes on day 1 of cycles 2-4. Patients also receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo lymphatic imaging with indocyanine green (ICG) prior to treatment start and blood sample collection throughout the study. (CLOSED TO ENROLLMENT)

COHORT B: Patients receive ipilimumab intra-lymphatically via DoseConnect™ and nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study and may optionally undergo lymphatic imaging with ICG prior to treatment start.

After completion of study treatment, patients are followed up every 4 months until disease progression, and then every 6 months for up to 2 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Measurable disease as defined below:

  * A non-nodal lesion is considered measurable if its longest diameter can be accurately measured as >= 2.0 cm with chest x-ray, or as >= 1.0 cm with computed tomography (CT) scan, CT component of a positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI)
  * A superficial non-nodal lesion is measurable if its longest diameter is >= 1.0 cm in diameter as assessed using calipers (e.g., skin nodules) or imaging. In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.
  * A malignant lymph node is considered measurable if its short axis is > 1.5 cm when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm).
  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease.
* Histologically or cytologically confirmed diagnosis of unresectable stage III or IV metastatic melanoma, meeting one of the following criteria:

  * Progressed after at least one line of FDA approved therapy [either immune checkpoint inhibitor (ICI) or targeted therapy]
  * Recurrent disease following initial surgical resection (may or may not have received adjuvant therapy)
  * Newly diagnosed or recurrent in-transit metastatic melanoma (may or may not be treatment naïve)
  * Progressed on at least one line of therapy containing anti-PD-1, antiPD-L1, or a BRAF inhibitor
* Hemoglobin >= 8.0 g/dL (obtained =< 15 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 15 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 15 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3.0 x ULN (obtained =< 15 days prior to registration)
* Serum creatinine =< 2.0 x ULN (obtained =< 15 days prior to registration)
* Calculated creatinine clearance >= 40 ml/min using the Cockcroft-Gault formula (obtained =< 15 days prior to registration)
* Prothrombin time (PT)/institutional normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy INR or aPTT is within target range of therapy (obtained =< 15 days prior to registration)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Persons able to become pregnant OR able to father a child must be willing to use an adequate method of contraception while on treatment and for 180 days (6 months) after last treatment dose on this study
* Provide written informed consent
* Patients enrolling in Rochester, Minnesota (MN), ONLY: Willingness to provide mandatory blood specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Metastatic sites that drain lymphatic fluid into nodal beds which are not amenable to lymphatic infusion

  * Sites of metastases limited only to the head and neck
  * Sites of metastatic disease limited to the lungs and/or hilar lymph nodes
* Metastatic uveal melanoma
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
  * Persons expecting to conceive or father children during the study or within 180 days (6 months) after the last treatment on this study
* Active central nervous system (CNS) metastases not previously treated

  * NOTE: patients with history of previously treated CNS metastases, not demonstrating evidence of progression for at least 12 weeks will be allowed
  * NOTE: patients with leptomeningeal metastases are not eligible
* Any of the following prior therapies:

  * Allogeneic hematopoietic stem cell transplantation (HSCT)
  * Solid organ transplantation
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Active autoimmune disease requiring systemic treatment < 2 years prior to registration, documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents with use of disease modifying agents, corticosteroids or immunosuppressive drugs. NOTE: Exceptions are allowed for the following conditions:

  * Vitiligo
  * Resolved childhood asthma/atopy
  * Intermittent use of bronchodilators or inhaled steroids
  * Daily steroids at dose of =< 10 mg of prednisone (or equivalent)
  * Local steroid injections
  * Stable hypothyroidism on replacement therapy
  * Stable diabetes mellitus on therapy (with or without insulin)
  * Sjogren's syndrome
  * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) which is not considered a form of systemic treatment and is allowed
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic therapy
  * Interstitial lung disease
  * Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
  * Known history of hepatitis B (i.e., known positive hepatitis B virus (HBV) surface antigen (HBsAg) reactive)
  * Known active hepatitis C (i.e., positive for hepatitis C virus (HCV) ribonucleic acid (RNA) detected by polymerase chain reaction (PCR))
  * Known active tuberculosis (TB)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia or
  * Psychiatric illness/social situations that would limit compliance with study requirements (e.g., known substance abuse)
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of severe hypersensitivity reactions to other monoclonal antibodies or known hypersensitivity to the study intervention or its excipients, indocyanine green (ICG) dye or iodine
* Prior history of grade 4 immune related adverse event (irAE) with prior intracavernosal injection (ICI) therapy or failure to recover (< grade 1) from immune-related adverse event(s) from prior ICI therapy
* Any of the following therapies prior to registration:

  * Chemotherapy =< 28 days
  * Immunotherapy =< 28 days
  * Targeted therapies (e.g., dabrafenib) =< 21 days
  * Other investigational agents =< 28 days
  * Radiation therapy =< 14 days
  * Minor surgical or interventional procedure =< 7 days
  * Major surgical procedure =< 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ipilimumab administration via the DoseConnect device in combination with nivolumab | Up to 21 days
  MTD is defined as the dose level where at most 1 of the 6 patients treated at that dose level develops a dose-limited event (DLE) during the first cycle of treatment and neither a Grade 3 or worse adverse event (AE) attributable to either drug or device or a Grade 2 or worse AE lasting ≥1 week and attributable to device reported after the first cycle of treatment.
Incidence of adverse events | Up to 21 days
  The maximum grade of each type of adverse event will be recorded for each patient. For each adverse event reported by dose level, the percentage of patients developing any degree of that adverse event as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.
Progression-free survival | Up to 2 years
  Defined as the time from study entry to the documentation of disease progression.
Overall survival | Up to 2 years
  Defined as the time from study entry to death.

OTHER OUTCOMES:
Immune parameter analysis | Up to 2 cycles (1 cycle = 21 days)
  For each individual, a time series plot of the fold increase in a given immune parameter from pre-treatment levels will be constructed to visual inspect for trends. An immune response in a given parameter will be defined as a two-fold or more increase from pre-treatment levels for those with detectable levels prior to treatment or a two-fold or more increase from the LLD for those with levels below the LLD prior to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Dimou, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States